CLINICAL TRIAL: NCT05836233
Title: Predictive Value of Vasodilator Challenge for Right Heart Failure (RHF) After Left Ventricular Assist Device (LVAD) Implantation
Brief Title: Predictive Value of Vasodilator Challenge for Right Heart Failure After LVAD Implantation
Acronym: PREVV-RHF-LVAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: San Camillo Hospital, Rome (Other)
Collaborators: Azienda Ospedaliero Universitaria, Santa Maria della Misericordia di Udine, Italy (Other)
Responsible Party: Principal Investigator, Giulio Cacioli, MD, San Camillo Hospital, Rome
Other Study IDs: 1235/CE Lazio 1
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Right Heart Failure
Keywords: LVAD; Right Heart Failure; Advanced Heart Failure; Nitroprusside; Right Heart Catheterization
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Enrolled patients - LVAD candidates: Inclusion criteria
  * Age over 18 years old.
  * Diagnosis of advanced heart failure with an indication for LVAD implantation.
  * Mean Arterial Pressure (MAP) > 60 mmHg; Mean Pulmonary Arterial Pressure (mPAP) > 20 mmHg; Pulmonary Artery Wedge Pressure >15 mmHg.
  * Vasodilator Challenge performed through NTP infusion.
  Exclusion criteria
  * State of pregnancy.
  * Inability to perform vasodilator challenge
  * Need for extracorporeal membrane oxygenator or short-term right ventricular assist devices.
  * Planned right ventricular assist device implantation in the peri-procedural setting.
  Interventions: Drug: Pulmonary Vasodilators

INTERVENTIONS:
Drug: Pulmonary Vasodilators — Right heart catheterization via Swan Ganz catether will be performed under optimal medical therapy within 90 days before LVAD implantation. We will record the timing between RHC and LVAD implantation.
  Vasodilator challenge will be performed through intravenous nitroprusside administration and titration (by 5 minutes intervals) until symptoms (flushing or hypotension) onset or systolic systemic pressure drop below 85 mmHg (target dose).
  Dobutamine or phosphodiesterase inhibitors infusion could be performed at clinician's discretion.
  All haemodynamic measurements will be repeated after nitroprusside infusion and titration until the target dose.
  Other Names: Vasodilator Challenge

SUMMARY:
Prospective evaluation of the predictive value for post-LVAD right ventricular failure (RHF) of pulmonary vasodilator challenge, in addition to current laboratory, echocardiographic and haemodynamic parameters.

LVAD candidates satisfying the inclusion criteria will undergo vasodilator challenge with sodium nitroprusside (NTP) infusion following the study protocol.

Thereafter, we will evaluate all data in order to determine which variables significantly correlate with RHF onset after LVAD implantation.

DETAILED DESCRIPTION:
Inclusion criteria

* Age over 18 years old.
* Diagnosis of advanced heart failure with an indication for LVAD implantation.
* Mean Arterial Pressure (MAP) > 60 mmHg; Mean Pulmonary Arterial Pressure (mPAP) > 20 mmHg; Pulmonary Artery Wedge Pressure >15 mmHg.
* Vasodilator Challenge performed through NTP infusion.

Exclusion criteria

* State of pregnancy.
* Inability to perform vasodilator challenge
* Need for extracorporeal membrane oxygenator or short-term right ventricular assist devices.
* Planned right ventricular assist device implantation in the peri-procedural setting.

Right heart catheterization (RHC) RHC will be performed under optimal medical therapy within 90 days before LVAD implantation.

Vasodilator challenge will be performed through intravenous nitroprusside administration and titration (by 5 minutes intervals) until symptoms (flushing or hypotension) onset or systolic systemic pressure drops below 85 mmHg.

Dobutamine or phosphodiesterase inhibitors infusion could be performed at clinician's discretion.

All haemodynamic measurements will be repeated after nitroprusside infusion and titration.

Right heart failure (RHF) Post-operative RHF will be evaluated according to the definition proposed by the 2020 consensus statement of the mechanical circulatory support academic research consortium (1).

ELIGIBILITY:
Inclusion criteria

* Age over 18 years old.
* Diagnosis of advanced heart failure with an indication for LVAD implantation.
* Mean Arterial Pressure (MAP) > 60 mmHg; Mean Pulmonary Arterial Pressure (mPAP) > 20 mmHg; Pulmonary Artery Wedge Pressure >15 mmHg.
* Vasodilator Challenge performed through NTP infusion.

Exclusion criteria

* State of pregnancy.
* Inability to perform vasodilator challenge
* Need for extracorporeal membrane oxygenator or short-term right ventricular assist devices.
* Planned right ventricular assist device implantation in the peri-procedural setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced heart failure patients undergoing left ventricular assist device implantation in our centers satisfying the inclusion criteria.
  All patients presenting one or more of the exclusion criteria will not be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 18 months
  Early right heart failure

SECONDARY OUTCOMES:
Secondary Endpoint | 24 months
  In-hospital all-cause mortality
Secondary Endpoint | 24 months
  1-year all-cause mortality;
Secondary Endpoint | 24 months
  Late right heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Musumeci, MD, Principal Investigator — San Camillo Hospital
Locations (1):
- San Camillo Hospital, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kormos RL, Antonides CFJ, Goldstein DJ, Cowger JA, Starling RC, Kirklin JK, Rame JE, Rosenthal D, Mooney ML, Caliskan K, Messe SR, Teuteberg JJ, Mohacsi P, Slaughter MS, Potapov EV, Rao V, Schima H, Stehlik J, Joseph S, Koenig SC, Pagani FD. Updated definitions of adverse events for trials and registries of mechanical circulatory support: A consensus statement of the mechanical circulatory support academic research consortium. J Heart Lung Transplant. 2020 Aug;39(8):735-750. doi: 10.1016/j.healun.2020.03.010. Epub 2020 Apr 18. No abstract available. PMID 32386998